CLINICAL TRIAL: NCT02945384
Title: Broader Implementation of a Successful Dual-Generation Intervention in Partnership With Head Start of Lane County
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 03172011.022
Record Dates: First submitted 2016-06-24; First posted 2016-10-26 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2019-04

CONDITIONS: School Readiness
Keywords: family well-being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Creating Connections (Experimental): Dual-generation intervention: child component delivered in classroom setting, parent component delivered in small-group setting
  Interventions: Behavioral: Creating Connections: Strong Families, Strong Brains
- Head Start as usual (No Intervention): Regular Head Start curriculum

INTERVENTIONS:
Behavioral: Creating Connections: Strong Families, Strong Brains — Dual-generation intervention
  Arms: Creating Connections

SUMMARY:
This project involves the development of a scaled-up model of a successful dual-generation intervention targeting attention, stress, and self-regulation in families attending Head Start, and improvements of outcome assessments of the intervention. The investigators hypothesize that families randomly assigned to receive the intervention, compared to families not receiving the intervention, will show improved brain function for attention and self-regulation and improved physiological function for stress regulation in both children and their parents, improvements in child school performance and cognition, and improvements in assessments of parent/family well being.

DETAILED DESCRIPTION:
Based on basic research on the neuroplasticity of attention, stress, and family dynamics, the investigators developed a successful dual-generation intervention that targets attention, stress, and self-regulation. The intervention has been shown to improve brain function for attention, cognition, and behavior in preschool children in Head Start (HS) and also improves communication skills and reduces stress in parents. This project involves the development of a scaled-up model of this intervention working with with Head Start of Lane County (HSOLC).

Goal 1: In partnership with HSOLC, the investigators have developed a scaled-up model of the intervention that is delivered by HS specialists and sustainable and replicable by other HS programs. This intervention is called Creating Connections: Strong Families, Strong Brains (CC).

Goal 2: To characterize the degree to which CC improves distal outcomes related to parent/family well-being by assessing health and safety outcomes in parents and children, parental education, financial literacy and decision making, household chaos, and biomarkers of allostatic load related to health outcomes.

Goal 3: To evaluate hypothesized mediating factors related to changes in family well-being, specifically changes in foundational systems (stress and self-regulation) by refining measures of family stress and self-regulation by assessing heart rate variability in parents and children and neurophysiological measures of self-regulation in parents.

Children and parents at randomly assigned HSOLC sites will receive CC, and other HSOLC sites will deliver the regular HS curriculum. The investigators hypothesize that participation in CC will result in improved brain function for attention and self-regulation as well as improved physiological function for stress regulation in both children and their parents compared to families not receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Student at Head Start of Lane County (child); parent of student at HSOLC (parent)

Exclusion Criteria:

* Not a native speaker of English or Spanish
* does not have normal hearing, vision, physical, motor, and emotional development
* has history of brain injury or disorder
* currently taking medications that affect brain function

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2800 (Estimated)
Dates: Start 2013-09; Primary Completion 2018-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Changes in brain function for selective attention: event-related potential (ERP) auditory selective attention paradigm (children and adults) | 3-6 months
  To measure brain function for selective attention using ERPs, participants selectively attend to one of two simultaneously presented stories that differ in location (left/right), voice (male/female), and content. ERPs are recorded to identical 100 msec probes embedded in stories when attended and unattended, and the effects of selective attention are quantified by comparing the brain response to probes embedded in the attended story with the response to identical probes embedded in the unattended story.
Changes in stress physiology: respiratory sinus arrhythmia (parasympathetic nervous system function) and pre-ejection period (sympathetic nervous system function) | 3-6 months
  RSA is an index of high-frequency beat-to-beat variability of the electrocardiogram (ECG) signal, while accounting for variability in respiration rate. PEP is the amount of time between depolarization of the left ventricle, seen in the ECG wave as the "Q" component directly preceding a heart beat, and subsequent ejection of blood through the ventricles, measured via the maximal rate of change in the impedance waveform of the subsequent "B" component. Baseline values of RSA and PEP will be acquired upon arrival to the lab during a five-minute neutral video of ocean scenes. Following this, RSA and PEP will be collected during two ERP paradigms measuring selective attention (children and adults) and self-regulation (adults only). After the tasks, physiology will be recorded during a final five-minute recovery period while a neutral video is shown.
Changes in child school performance: Head Start Teaching Strategies Gold assessments | 3-6 months
Changes in child behavior for cognition: language (Clinical Evaluation of Language Fundamentals-Preschool: 2nd Ed.), IQ (Stanford-Binet Intelligence Scales-5th Ed.), executive function (Snack Delay, Shape School, Noisy Book) | 3-6 months
Changes in brain function for self-regulation: event-related potential (ERP) stop-signal task paradigm (adults only) | 3-6 months
  Brain function for self-regulation will be measured with an ERP variant of the stop-signal task with an added feedback component. Each trial begins with a fixation cross for 500 ms, followed by an arrow cue pointing either left or right for 500 ms (the "go signal"), a feedback stimulus presented 400-600 ms after a response and remaining on the screen for 100 ms, and finally a jittered intertrial interval of 2000 to 4000 ms. On 25% of trials, an auditory stop signal is played at a variable latency and adjusts trial-by-trial to appear 50 ms earlier following failed stops and 50 ms later after successful stops, while adjusting to maintain 50% response accuracy over blocks of eight stop trials. Shorter delay between cue and stop signal for successful stops indicates better inhibitory control. ERPs will be averaged to the onset of auditory stop signals, responses, and feedback stimuli.

SECONDARY OUTCOMES:
Changes in child social behavior: Preschool and Kindergarten Behavior Scale - 2nd Ed. | 3-6 months
Changes in parenting behavior: videotaped parent-child interactions coded for parent language behavior using Systematic Analysis of Language Transcripts-8 | 3-6 months
Changes in parenting stress: Parenting Stress Index | 3-6 months
Changes in home environment: Confusion, Hubbub, and Order Scale (CHAOS) | 3-6 months
Changes in adult health: systolic and diastolic blood pressure | 3-18 months
Changes in family well-being: Head Start Family Partnership Plan (FPP): Assessment of Strengths, Capabilities, & Needs | 3-18 months
Changes in home environment: Tayside Children's Sleep Questionnaire | 3-6 months
Changes in adult health: blood spot biomarkers of immune function | 3-18 months
  Immune function will be assessed via the following biomarkers: C-reactive protein, Epstein-Barr Virus antibodies, interleukin-6
Changes in adult health: blood spot biomarkers metabolic function | 3-18 months
  Metabolic function will be assessed via the following biomarkers: insulin, glycosylated hemoglobin (hemoglobin A1c) lipoprotein(a)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pakulak, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

REFERENCES:
- [Background] Neville HJ, Stevens C, Pakulak E, Bell TA, Fanning J, Klein S, Isbell E. Family-based training program improves brain function, cognition, and behavior in lower socioeconomic status preschoolers. Proc Natl Acad Sci U S A. 2013 Jul 16;110(29):12138-43. doi: 10.1073/pnas.1304437110. Epub 2013 Jul 1. PMID 23818591